CLINICAL TRIAL: NCT06135428
Title: The Effect of Training Based on the Midwifery Resilience Model on the Resilience of Midwives: Randomized Controlled Trial
Brief Title: The Effect of Training Based on the Midwifery Resilience Model
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Amasya University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: AmasyaTez
Record Dates: First submitted 2023-11-13; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Midwifery
Keywords: midwifery; training programs; resistance
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Training content was prepared in three stages according to the "resilience model in midwives". The training will be in the form of 45-minute presentations and sharings, and individual studies will be carried out in the form of homework according to people's methods of coping with stress. These homework assignments may occasionally include more or less individual meetings depending on the person's coping situation. However, at least 3 meetings will be held. Training and interviews will be conducted by researchers. For this, at least one of the researchers will receive training including personal awareness and motivational interviews.
  Interventions: Other: Education Group
- Control (No Intervention): No intervention

INTERVENTIONS:
Other: Education Group — Training content was prepared in three stages according to the "resilience model in midwives". The training will be in the form of 45-minute presentations and sharings, and individual studies will be carried out in the form of homework according to people's methods of coping with stress. These homework assignments may occasionally include more or less individual meetings depending on the person's coping situation. However, at least 3 meetings will be held. Training and interviews will be conducted by researchers. For this, at least one of the researchers will receive training including personal awareness and motivational interviews.
  Other Names: Control Group
  Arms: Experimental

SUMMARY:
Midwives' busy working environments, long working hours, worry of being sued, and encountering problems that may cause trauma can negatively affect their psychological resilience by increasing the stress level of midwives (Yalçın D., Bürün Bingöl F., 2023). Resilience in midwifery is a less researched topic (Sayıner F.D., Çömezoğlu E. et al., 2021). In studies investigating resilience in midwifery; Midwives' secondary traumatic stress total score was found to be high, while their resilience scale total score was found to be low. A negative, highly and statistically significant relationship was detected between the secondary traumatic stress scale and psychological resilience scale scores (r=-0.752; p=0.000) (Dağlı E., Topkara F.N., 2023). In another study, the factors affecting midwives' intention to change jobs or leave the profession were investigated. As a result; It was determined that almost half of the midwives intended to change jobs and/or quit midwifery within 5 years, and the most common reasons for the intention to change jobs/leave were family commitments, working conditions, role dissatisfaction, work-life balance and career change (Pugh J.D., 2013). So, it is recommended to develop programs to increase their quality of life and psychological resilience and to demonstrate their effectiveness through experimental studies (Sevin B., Partlak Gunüşen N., 2021).

Hypotheses:

H0. Training given according to the "midwifery resilience model" does not change midwives' resilience scale scores.

H1: Training given according to the "midwifery resilience model" increases midwives' resilience scale scores.

DETAILED DESCRIPTION:
Study Design The research is of the pre-test post-test randomized controlled experimental design type.

Details of Working Method 200 midwives working in Amasya public hospitals constitute the population of the research. The number of samples was calculated using the G.Power 3.1.9.4 analysis program. According to the one-way independent samples t test analysis with 95% confidence (1-α), 80% test power (1-β) and d = 0.5 effect size, the number of samples to be taken in each group was determined as 51. Considering that there may be losses in the number of samples, it is planned to take 10% more than the number of samples and make a total of 112 people, 56 people for each group. People who agree to participate in the research will be divided into two groups, the training group and the control group, using a computer-based randomization program (https://www.random.org/).

APPLICATION:

After the training group and control group are created, data collection forms (Appendix 1,2,3) will be applied to both groups.

After the pretests are administered, training will begin for the training group, and no intervention will be made to the control group. Immediately after the training is completed and 1 month later, the adult resilience scale and perceived stress scale will be filled in again in both groups.

Educational Intervention:

Training content was prepared in three stages according to the "resilience model in midwives". The training will be in the form of 45-minute presentations and sharings, and individual studies will be carried out in the form of homework according to people's methods of coping with stress. These homework assignments may occasionally include more or less individual meetings depending on the person's coping situation. However, at least 3 meetings will be held. Training and interviews will be conducted by researchers. For this, at least one of the researchers will receive training including personal awareness and motivational interviews.

Educational content:

Training Content, Hunter et al. It was prepared according to the midwifery resilience model he developed. There are 3 stages in this model. These; They are personal awareness, sensitive strategies and proactive strategies (8).

1. Self-Awareness Developing personal awareness includes knowing oneself, establishing realistic expectations, and developing a strong professional identity.

Self-Knowing of People; Self-knowledge is the basis of healthy communication and empathy (Karaca S., 2010). A person who knows himself is aware of both the external world and the internal world. Thus, a person can easily direct his own life (Cüceloğlu D., 1998). Self-knowledge begins with the family and is also affected by the culture (Burger JM., 2006). Self-awareness means knowing one's strengths, weaknesses, aspects that are open to improvement, and feelings, and using this awareness to guide thoughts and behaviors, and being able to express oneself clearly (Üstün B., Akgün E., Partlak N., 2005).

Self-knowledge occurs in 4 dimensions;

1. Psychological dimension; It is recognizing a person's emotions, thoughts, situations that affect them, and their personality.
2. Physical size; It is a person's body image and knowing himself physically.
3. Social dimension; It is the communication that a person establishes with other people.
4. Philosophical dimension; It is recognizing people's life, values and beliefs (Terakye G., 1995).

Realistic expectations; Be aware of your own needs and abilities. Avoid unrealistic expectations of both yourself and others (Sayıner F.D., Çömezoğlu E. et al., 2021).

Develop a strong professional identity; Having a strong professional identity and love for your profession can strengthen you in difficult times. Remember the importance of yourself and the people you care for in such difficult times (Sayıner F.D., Çömezoğlu E. et al., 2021).

2. Responsive strategies It includes developing ways to create positive moods, such as accessing social support, music and exercise, and trying to maintain work-life balance.

Access to social support; Social support is the foundation of resilience. Get support from your close friends and colleagues and chat with them (Sayıner F.D., Çömezoğlu E. et al., 2021). If you have a knowledgeable, experienced and supportive person who can give you perspective and support, especially in difficult situations, you can also get help from them. Apart from this, the support of family members is also important (Hunter B., Warren L., 2013).

Positive mood creation, such as music and exercise; You can do various activities to improve your mood. These; Going out, walking, exercising, or pursuing a hobby if you have one. At the same time, listening to music and taking a shower will relax you (Sayıner F.D., Çömezoğlu E. et al., 2021). You can talk about other topics, and you can reassure yourself in difficult or stressful situations by thinking that it will end (Hunter B., Warren L., 2013).

Developing ways to try to maintain work-life balance; Try to keep work and home life separate. Something that is good for you outside of work.

Data will be collected through face-to-face interviews with midwives who agreed to participate in the study. In the study, data will be collected from midwives using the Personal Information Form (Appendix-1), Psychological Resilience Scale for Adults (Appendix-2) and Perceived Stress Scale (Appendix-3).

1. Personal Information Form:

   The personal information form consists of a total of 23 questions, which include information about sociodemographic (age, marital status, education level, number of children), midwifery profession, and problems related to working conditions, after examining the literature by the researchers.
2. Psychological Resilience Scale for Adults:

The Psychological Resilience Scale for Adults, consisting of 33 items, was developed by Friborg et al. (2003) and includes the dimensions of 'personal strength', 'structural style', social competence', 'family harmony' and 'social resources'. A later study showed that the scale better explains the psychological resilience model with its six-dimensional structure. The Turkish validity and reliability study of the scale was conducted by Basım and Çetin (2011). Cronbach's alpha value was found to be 0.74. It has been reported that the Psychological Resilience Scale for Adults, adapted into Turkish, is reliable and valid at psychometrically acceptable levels (Basım H.N, Çetin F., 2011). 3.Perceived Stress Scale:

Perceived Stress Scale (PSS) was developed by Cohen, Kamarck and Mermelstein (1983). ASQ, consisting of a total of 14 items, is designed to measure how stressful some situations in a person's life are perceived. Participants evaluate each item on a 5-point Likert-type scale ranging from "Never (0)" to "Very often (4)". 7 of the items containing positive statements are reverse scored. In addition to the fourteen-item long form, ASQ has two other forms: 10 and 4-item. In this study, the reliability and validity of all three forms are tested. ASQ items (reverse scored items and items forming the 10- and 4-item form are also marked) are given in ANNEX-3. While the scores of ASÖ-14 vary between 0 and 56, the scores of ASÖ-10 vary between 0 and 40, and the scores of ASÖ-4 vary between 0 and 16. A high score indicates a person's perception of stress is high. The adaptation of this scale into Turkish and its reliability and validity analysis were conducted by Eskin M. et al. in 2013. Cronbach's alpha value was found to be 0.84. The findings obtained from this study show that the ASQ items have sufficient internal consistency and test-retest reliability. Additionally, the findings reveal that the PSS consists of two factors, self-efficacy and stress perception, and is a measurement tool with a high level of concurrent validity. Considering the findings of the study, the long and short forms of the Turkish ASQ can be used as a valid and reliable measurement tool to measure people's perceptions of stress in their lives (Eskin M. et al., 2013).

* Inclusion Criteria
* Midwives who agreed to participate in the study.
* Statistical Methods
* Stastical Package for Social Science for Windows SPSS package program will be used to analyze the data. In data analysis, ordinal variables will be evaluated as arithmetic mean and standard deviation, minimum and maximum. As statistical analysis methods, Student's t test and one-way variance (One Way ANOVA), the relationship will be examined with Pearson Product Moment Correlation Coefficient and Mann-Whitney U test, and the significance level will be evaluated as p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Midwives who agreed to participate in the study.

Exclusion Criteria:

-

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2023-12-20 (Estimated); Study Completion 2024-02-10 (Estimated)

PRIMARY OUTCOMES:
Scale-1 | immediately after training
  Psychological Resilience Scale for Adults
Scale-2 | immediately after training
  Perceived Stress Scale

SECONDARY OUTCOMES:
Scale-1 | one month after the unit of training
  Psychological Resilience Scale for Adults
Scale-2 | one month after the unit of training
  Perceived Stress Scale

CONTACTS AND LOCATIONS:
Overall Officials: Duygu Murat Öztürk, Study Director — Amasya üniversitesi
Locations (1):
- Amasya University Faculty of Health Sciences, Amasya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lopes SC, Titulaer P, Bokosi M, Homer CS, ten Hoope-Bender P. The involvement of midwives' associations in policy and planning about the midwifery workforce: A global survey. Midwifery. 2015 Nov;31(11):1096-103. doi: 10.1016/j.midw.2015.07.010. Epub 2015 Jul 29. PMID 26304303
- [Result] Crowther S, Hunter B, McAra-Couper J, Warren L, Gilkison A, Hunter M, Fielder A, Kirkham M. Sustainability and resilience in midwifery: A discussion paper. Midwifery. 2016 Sep;40:40-8. doi: 10.1016/j.midw.2016.06.005. Epub 2016 Jun 8. PMID 27428097
- [Result] Hunter B, Warren L. Midwives׳ experiences of workplace resilience. Midwifery. 2014 Aug;30(8):926-34. doi: 10.1016/j.midw.2014.03.010. Epub 2014 Mar 26. PMID 24742637
- [Result] Pugh JD, Twigg DE, Martin TL, Rai T. Western Australia facing critical losses in its midwifery workforce: a survey of midwives' intentions. Midwifery. 2013 May;29(5):497-505. doi: 10.1016/j.midw.2012.04.006. Epub 2012 Nov 22. PMID 23182501
- [Derived] Hacikoylu E, Murat Ozturk D. The effect of educational intervention based on midwifery resilience model on midwives' resilience and stress levels: a randomized controlled trial. BMC Nurs. 2025 Jun 3;24(1):629. doi: 10.1186/s12912-025-03298-0. PMID 40462056